CLINICAL TRIAL: NCT01269021
Title: Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, China.
Brief Title: An Multi-site Prospective Study to Assess the Efficacy and Safety of MMF in the Treatment of Proliferative IgA Nephropathy(IgAN)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Zhi-Hong Liu, M.D. (Other)
Responsible Party: Sponsor-Investigator, Zhi-Hong Liu, M.D., professor, Nanjing University School of Medicine
Organization: Nanjing University School of Medicine (Other)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: NJCT-1005
Record Dates: First submitted 2010-12-10; First posted 2011-01-04 (Estimated); Last update posted 2016-03-17 (Estimated); Status verified 2016-03

CONDITIONS: IgA Nephropathy (IgAN)
Keywords: MMF treatment IgA Nephropathy (IgAN)
MeSH Terms: conditions — Glomerulonephritis, IGA | interventions — Mycophenolic Acid; Prednisone

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- mycophenolate mofetil (Experimental)
  Interventions: Drug: mycophenolate mofetil plus lower dose of Prednisone
- Prednisone (Active Comparator)
  Interventions: Drug: Prednisone in full dose

INTERVENTIONS:
Drug: mycophenolate mofetil plus lower dose of Prednisone — MMF 1.0-1.5g/d*6mons Prednisone 0.4-0.6 mg/kg/d
  Other Names: MMF
  Arms: mycophenolate mofetil
Drug: Prednisone in full dose — 0.8-1mg/kg/d
  Arms: Prednisone

SUMMARY:
In order to treat proliferative IgA Nephropathy(IgAN), The investigators designed an open, prospective, randomized parallel study to access the efficacy and safety of MMF compared to corticosteroid .

Patients who fulfill the inclusion criteria will be randomized in a 1:1 ratio to either the MMF group or corticosteroid group.

DETAILED DESCRIPTION:
To access the efficacy and safety of MMF compared to corticosteroid in in treatment of proliferative IgA Nephropathy(IgAN).

ELIGIBILITY:
Inclusion Criteria:

1. Patients who signed written informed consent form
2. age between 18-60 years, female or male
3. diagnosed IgA Nephropathy (IgAN) by renal biopsy during 1 months
4. renal biopsy had: 10%< crescents<50%; endocapillary hypercellularity; or necrosis ,and interstitial fibrosis<50%,
5. proteinuria>1g/24h for two times

Exclusion Criteria:

1. secondary IgA Nephropathy (IgAN);
2. eGFR<30ml/min/1.73m2.( MDRD formula)
3. liver disfunction;
4. uncontrolled hypertension
5. WBC <3000/mm3
6. Severe viral infection(HBV, HCV, CMV) within 3 months ofor known HIV infection.
7. diabetes or obesity(BMI>28) ;
8. severe infection or central nervous system symptoms.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 176 (Actual)
Dates: Start 2010-11; Primary Completion 2013-10 (Actual); Study Completion 2014-04 (Actual)

PRIMARY OUTCOMES:
the rate of complete remission (CR) at 6 months | 6 months

SECONDARY OUTCOMES:
the rate of overall response (CR+ partial remission [PR]) at 6 months | 6 months
the median time to CR | from the start of enrollment to the day of complete remission
the relapse rate after stopping the treatments | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Zhihong Liu, Master, Principal Investigator — Research Institute of Nephrology, Jinling Hospital, Nanjing University School of Medicine, Nanjing, China.
Locations (1):
- Research Institute of Nephrology, Nanjing, Jiangsu, China